CLINICAL TRIAL: NCT05327088
Title: Effect of Epidural Dexmedetomidine VS Nalbuphine for Labor Analgesia
Brief Title: Epidural Dexmedetomidine vs Nalbuphine for Labor Analgesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nourhan Tarek, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Epidural analgesia
Record Dates: First submitted 2022-03-28; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Epidural Anesthesia; Labor Pain
Keywords: Dexmedetomidine; Nalbuphine
MeSH Terms: conditions — Labor Pain | interventions — Dexmedetomidine; Nalbuphine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Dexmedetomidine group) (Active Comparator): a bolus dose of 11ml of 0.25% bupivacaine + 0.5μg/ml preservative free dexmedetomidine (1ml volume) will be injected via the epidural catheter. For top up 5 ml of 0.25% bupivacaine + 0.5μg/ml dexmedetomidine (1ml volume) will be given when VAS score becomes 4 or more.
  Interventions: Drug: Dexmedetomidine
- Group B (Nalbuphine group) (Active Comparator): a bolus dose of 11ml of 0.25% bupivacaine + 10mg preservative free nalbuphine (1ml volume) will be injected via the epidural catheter. For top up 5 ml of 0.25% bupivacaine + 2mg nalbuphine (1ml volume) will be given when VAS score becomes 4 or more.
  Interventions: Drug: Nalbuphine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine, a highly selective α₂ receptor agonist, has a sympatholytic, sedative and opioid sparing effect.
  Other Names: Precedex
  Arms: Group A (Dexmedetomidine group)
Drug: Nalbuphine — Nalbuphine, a derivative of 14-hydroxymorphine is a strong analgesic with mixed k agonist and µ antagonist properties. The analgesic potency of nalbuphine has been found to be equal to morphine
  Other Names: Nalufin
  Arms: Group B (Nalbuphine group)

SUMMARY:
The aim of this study is to compare epidural dexmedetomidine vs nalbuphine added to bupivacaine in labor analgesia and determine the privilege of one over the other and to compare the effect of both analgesics after delivery.

DETAILED DESCRIPTION:
Labor pain often causes a strong stress response in women. Recently, it is concerned by most mothers and doctors that how to effectively alleviate the pain during delivery. There is no standard treatment for labor pain. A wide range of pharmacological and non-pharmacological labor pain relief techniques are available for pregnant women . Labor analgesia, also known as painless childbirth, refers to the use of various methods to reduce maternal labor pain or make it disappear. The ideal labor analgesia should be based on maternal and child safety, and should have fast acting, good analgesic effect and less adverse reaction. Epidural block anesthesia is convenient, and has less adverse reaction and obvious effect in the commonly used analgesic methods, which is widely used in the current way of analgesia. Dexmedetomidine is a highly selective α2 adrenergic receptor agonist that has sedative, hypnotic, and analgesic effects . Nalbuphine is a synthetic agonist antagoLabor pain often causes a strong stress response in women. Recently, it is concerned by most mothers and doctors that how to effectively alleviate the pain during delivery. There is no standard treatment for labor pain. A wide range of pharmacological and non-pharmacological labor pain relief techniques are available for pregnant women . Labor analgesia, also known as painless childbirth, refers to the use of various methods to reduce maternal labor pain or make it disappear. The ideal labor analgesia should be based on maternal and child safety, and should have fast acting, good analgesic effect and less adverse reaction. Epidural block anesthesia is convenient, and has less adverse reaction and obvious effect in the commonly used analgesic methods, which is widely used in the current way of analgesia. Dexmedetomidine is a highly selective α2 adrenergic receptor agonist that has sedative, hypnotic, and analgesic effects . Nalbuphine is a synthetic agonist antagonist opioid that has the characteristics of mu-antagonist and kappa-agonist activities. Nalbuphine has gained popularity as a parenteral analgesic for intraoperative, postoperative, and obstetrical uses . The purpose of this study is to compare between the 2 drugs in decreasing labor pain. st opioid that has the characteristics of mu-antagonist and kappa-agonist activities. Nalbuphine has gained popularity as a parenteral analgesic for intraoperative, postoperative, and obstetrical uses . The purpose of this study is to compare between the 2 drugs in decreasing labor pain.

ELIGIBILITY:
Inclusion Criteria:

All the parturients should :

1. Be between 21 - 40 years old
2. ASA classification I- II
3. Para 1-2
4. Requesting analgesia
5. Have a normal birth canal
6. Be at the beginning of active phase of labor i.e. cervical dilatation of 4 cm with regular uterine contractions.
7. The fetus should be a single full-term fetus (37- 42 weeks of gestation) with normal head position, normal development.

Exclusion Criteria:

Parturients

1. Younger than 21 and older than 40 years old
2. With contraindication of regional anesthesia
3. With pre-existing neurological disease
4. With history of allergy to the study drugs
5. With cephalopelvic disproportion, fetal distress, amniotic fluid infection, placental insufficiency or scarred uterus

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2021-09-12 (Actual); Primary Completion 2022-02-12 (Actual); Study Completion 2022-03-12 (Actual)

PRIMARY OUTCOMES:
change in VAS score for pain before analgesia and every 30 minutes after analgesia | before analgesia and 30 minutes after analgesia and then every 30 minute as long as the epidural catheter is inserted (up to 360 minutes)
  The visual analog scale (VAS) is a tool widely used to measure pain. A patient is asked to indicate his/her perceived pain intensity along a 100 mm (10 cm) horizontal line, and this rating is then measured from the left edge (=VAS score). The VAS score correlates well with acute pain levels (Myles et al., 1999). Using a ruler, the score is determined by measuring the distance (cm) on the 10-cm line between the no pain anchor and the patients mark, providing a range of scores from 010. A higher score indicates greater pain intensity.

SECONDARY OUTCOMES:
change in Heart rate before analgesia and every 30 minutes after analgesia | before analgesia and 30 minutes after analgesia and then every 30 minute as long as the epidural catheter is inserted (up to 360 minutes)
  Monitored and recorded
change in arterial blood pressure before analgesia and every 30 minutes after analgesia | before analgesia and 30 minutes after analgesia and then every 30 minute as long as the epidural catheter is inserted (up to 360 minutes)
  Monitored and recorded
change in SpO2 before analgesia and every 30 minutes after analgesia | before analgesia and 30 minutes after analgesia and then every 30 minute as long as the epidural catheter is inserted (up to 360 minutes)
  Monitored and recorded
Duration of active phase of 1st stage of labor | from 100 minutes to 300 minutes
  The duration of active phase of 1st stage of labor varies from one to the other
Duration of 2nd stage of labor | from 30 minutes to 200 minutes
  The duration of 2nd stage of labor varies from one to the other
Duration of 3rd stage of labor | from 5 minutes to 15 minutes
  The duration of 3rd stage of labor varies from one to the other
Neonatal condition: APGAR score at 1 and 5 min after the birth | At 1 minute and 5 minutes after birth
  to check if any of the study drugs can deteriorate the neonatal condition
The adverse reactions: itching, nausea, vomiting, bradycardia and hypotension | As long as the epidural catheter is inserted (up to 360 minutes)
  These adverse reaction can occur after administration of the interventional drugs

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

REFERENCES:
- [Background] Abdalla W, Ammar MA, Tharwat AI. Combination of dexmedetomidine and remifentanil for labor analgesia: A double-blinded, randomized, controlled study. Saudi J Anaesth. 2015 Oct-Dec;9(4):433-8. doi: 10.4103/1658-354X.159470. PMID 26543463
- [Background] Camann WR, Hurley RH, Gilbertson LI, Long ML, Datta S. Epidural nalbuphine for analgesia following caesarean delivery: dose-response and effect of local anaesthetic choice. Can J Anaesth. 1991 Sep;38(6):728-32. doi: 10.1007/BF03008450. PMID 1914055
- [Background] Chatrath V, Attri JP, Bala A, Khetarpal R, Ahuja D, Kaur S. Epidural nalbuphine for postoperative analgesia in orthopedic surgery. Anesth Essays Res. 2015 Sep-Dec;9(3):326-30. doi: 10.4103/0259-1162.158004. PMID 26712968
- [Background] Czech I, Fuchs P, Fuchs A, Lorek M, Tobolska-Lorek D, Drosdzol-Cop A, Sikora J. Pharmacological and Non-Pharmacological Methods of Labour Pain Relief-Establishment of Effectiveness and Comparison. Int J Environ Res Public Health. 2018 Dec 9;15(12):2792. doi: 10.3390/ijerph15122792. PMID 30544878
- [Background] Aveline C, Bonnet F. [The effects of peridural anesthesia on duration of labor and mode of delivery]. Ann Fr Anesth Reanim. 2001 May;20(5):471-84. doi: 10.1016/s0750-7658(01)00398-7. French. PMID 11419241
- [Background] Li N, Hu L, Li C, Pan X, Tang Y. Effect of Epidural Dexmedetomidine as an Adjuvant to Local Anesthetics for Labor Analgesia: A Meta-Analysis of Randomized Controlled Trials. Evid Based Complement Alternat Med. 2021 Oct 27;2021:4886970. doi: 10.1155/2021/4886970. eCollection 2021. PMID 34745286
- [Background] Wangping Z, Ming R. Optimal Dose of Epidural Dexmedetomidine Added to Ropivacaine for Epidural Labor Analgesia: A Pilot Study. Evid Based Complement Alternat Med. 2017;2017:7924148. doi: 10.1155/2017/7924148. Epub 2017 Jun 1. PMID 28656055